CLINICAL TRIAL: NCT00134316
Title: Cervical or Endometrial Cancer and Sexual Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Lori Brotto, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBC-SH-CECSH.P1&2-20R91396; CIHR-PG#20R91396
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Sexual Dysfunctions, Psychological
Keywords: sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: psychoeducational intervention — three 75 minute long individual psychoeducational sessions

SUMMARY:
Aim #1. To investigate the efficacy of the psychoeducational intervention (PED) on sexual arousal.

H1: Compared to a control group and to baseline, PED will result in significant improvement in:

* self-reported subjective sexual arousal;
* self-reported genital sensitivity;
* psychophysiological sexual arousal.

Aim #2. To investigate the efficacy of the PED on self-reported orgasm, sexual desire, distress, and relationship satisfaction.

H2: Compared to a control group and to baseline, PED will result in significant improvement in self-reported orgasmic experience, sexual desire, sexual distress, and relationship satisfaction.

Aim #3. To investigate the efficacy of the PED on depressive symptoms and quality of life.

H3: Compared to a control group and to baseline, PED will result in significant improvement in self-reported depressive symptoms and quality of life.

DETAILED DESCRIPTION:
Whereas relatively more research and therapy options exist for physical treatments of sexual dysfunction in women with a history of cervical cancer (e.g. hormone replacement, surgery; Denton & Maher, 2003), there is some evidence that psychological interventions have positive effects on sexuality. For example, a brief psychoeducational program for women with early-stage cervical cancer resulted in significant improvements in the frequency of coital activity (Capone et al., 1980), and enhanced compliance with sexual rehabilitation, reduced fear about intercourse and improved sexual knowledge compared to a control condition (Robinson et al., 1999). Unfortunately, neither study targeted nor assessed sexual arousal or genital sensations - symptoms documented to be most problematic and distressing in this group of women. There is also evidence that providing a venue for women to receive education and discuss sexual concerns following cervical cancer is therapeutic as it might encourage women to be more aware of their sexual rehabilitation and capacity for change, thus evoking a more active coping style (Leenhouts et al., 2002). Taken together, these studies suggest that psychoeducational interventions are feasible and significantly improve general domains of sexual function, such as sexual frequency and knowledge, in cervical cancer survivors.

Although directly targeting psychological constructs such as thoughts, affect, and behaviour, psychological treatments can also evoke physiological change. In cervical cancer-related sexual dysfunction where the psychological and physical contributors of impairment are difficult to tease apart, a psychoeducational intervention that addresses both etiological domains is essential. We have recently developed a 3-session psychoeducational intervention designed to address both the physical and psychological consequences of cervical cancer on sexual arousal. The sexual arousal concerns reported by this group of women fit the criteria for Female Sexual Arousal Disorder (FSAD), defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revised (DSM-IV-TR) as "persistent or recurrent inability to attain, or to maintain until completion of the sexual activity, an adequate lubrication-swelling response of sexual excitement" where "the disturbance causes marked distress or interpersonal difficulty" (American Psychiatric Association, 2000). A proportion of these women also experience new onset difficulties becoming subjectively sexually aroused, likely as a direct result of the genital arousal difficulties, but also due to the impact of cancer and hysterectomy on psychological function. Despite the wide prevalence of such subjective arousal concerns, this is not a diagnostic category in the DSM-IV-TR. However, the International Consultation on Sexual Dysfunctions, in collaboration with the World Health Organization, has suggested that "Subjective Sexual Arousal Disorder" be recognized as a valid concern (Basson et al., 2003). Evidence-based treatments for FSAD related to genital or subjective arousal difficulties do not exist, and persisting distress due to untreated sexual dysfunction can compromise mental and physical health. The contents of our psychoeducational intervention were based on:

* empirically supported techniques in other areas of female sexual dysfunction (e.g., sensate focus, challenging of maladaptive cognitions and sexual myths);
* discussions with gynecological oncologists at the University of Washington who are usually the first-line recipients of such sexual complaints; and
* pilot interviews conducted with 18 cervical and endometrial cancer survivors to date.

The intervention focuses primarily on sexual arousal, both genital and subjective, and secondarily on the interaction between cervical cancer and hysterectomy with relationship satisfaction, body image, and beliefs about health.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervical or endometrial cancer, in remission for at least 1 year
* Treatment by hysterectomy at least one year earlier
* Diagnosis of female sexual arousal disorder (FSAD) according to DSM-IV-TR criteria with new onset after the hysterectomy
* Currently involved in a relationship

Exclusion Criteria:

* Treatment by either radiation or chemotherapy alone
* Current diagnosis of primary hypoactive sexual desire disorder - or in other words, if complaints of sexual desire are present, they must be less distressing than the sexual arousal complaints.
* Unstable psychopathology and Beck Depression Inventory scores greater than 19
* Lack of sexual experience
* Current use of antidepressants or other medication with known sexual side effects
* Those with a physical condition that would impede participation in the psychophysiological assessment

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-08; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Upon completion of data analysis, establishment of the efficacy of a psychoeducational intervention (PED) in a sample of cervical or endometrial cancer survivors with sexual arousal disorder will be determined. | upon completion of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Basson, FCRP (UK), Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Butler L, Banfield V, Sveinson T, Allen K. Conceptualizing sexual health in cancer care. West J Nurs Res. 1998 Dec;20(6):683-99; discussion 700-5. doi: 10.1177/019394599802000603. PMID 9842287
- [Background] Butler-Manuel SA, Buttery LD, A'Hern RP, Polak JM, Barton DP. Pelvic nerve plexus trauma at radical and simple hysterectomy: a quantitative study of nerve types in the uterine supporting ligaments. J Soc Gynecol Investig. 2002 Jan-Feb;9(1):47-56. doi: 10.1016/s1071-5576(01)00145-9. PMID 11839509
- [Background] Grumann M, Robertson R, Hacker NF, Sommer G. Sexual functioning in patients following radical hysterectomy for stage IB cancer of the cervix. Int J Gynecol Cancer. 2001 Sep-Oct;11(5):372-80. doi: 10.1046/j.1525-1438.2001.01051.x. PMID 11737468
- [Background] Juraskova I, Butow P, Robertson R, Sharpe L, McLeod C, Hacker N. Post-treatment sexual adjustment following cervical and endometrial cancer: a qualitative insight. Psychooncology. 2003 Apr-May;12(3):267-79. doi: 10.1002/pon.639. PMID 12673810
- [Background] Kylstra WA, Leenhouts GH, Everaerd W, Panneman MJ, Hahn DE, Weijmar Schultz WC, Van De Wiel HB, Heintz AP. Sexual outcomes following treatment for early stage gynecological cancer: a prospective multicenter study. Int J Gynecol Cancer. 1999 Sep;9(5):387-395. doi: 10.1046/j.1525-1438.1999.99052.x. PMID 11240799
- [Background] Robinson JW, Faris PD, Scott CB. Psychoeducational group increases vaginal dilation for younger women and reduces sexual fears for women of all ages with gynecological carcinoma treated with radiotherapy. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):497-506. doi: 10.1016/s0360-3016(99)00048-6. PMID 10348277
- [Background] Wenzel LB, Donnelly JP, Fowler JM, Habbal R, Taylor TH, Aziz N, Cella D. Resilience, reflection, and residual stress in ovarian cancer survivorship: a gynecologic oncology group study. Psychooncology. 2002 Mar-Apr;11(2):142-53. doi: 10.1002/pon.567. PMID 11921330
- [Background] Andersen BL, Woods XA, Copeland LJ. Sexual self-schema and sexual morbidity among gynecologic cancer survivors. J Consult Clin Psychol. 1997 Apr;65(2):221-9. doi: 10.1037//0022-006x.65.2.221. PMID 9086685
- [Background] Anderson BJ, Wolf FM. Chronic physical illness and sexual behavior: psychological issues. J Consult Clin Psychol. 1986 Apr;54(2):168-75. doi: 10.1037//0022-006x.54.2.168. No abstract available. PMID 3700803
- [Background] Butler-Manuel SA, Buttery LD, A'Hern RP, Polak JM, Barton DP. Pelvic nerve plexus trauma at radical hysterectomy and simple hysterectomy: the nerve content of the uterine supporting ligaments. Cancer. 2000 Aug 15;89(4):834-41. doi: 10.1002/1097-0142(20000815)89:43.0.co;2-7. PMID 10951347
- [Background] Capone MA, Good RS, Westie KS, Jacobson AF. Psychosocial rehabilitation of gynecologic oncology patients. Arch Phys Med Rehabil. 1980 Mar;61(3):128-32. PMID 7369850
- [Background] Leenhouts GH, Kylstra WA, Everaerd W, Hahn DE, Schultz WC, van de Wiel HB, Heintz AP. Sexual outcomes following treatment for early-stage gynecological cancer: a prospective and cross-sectional multi-center study. J Psychosom Obstet Gynaecol. 2002 Jun;23(2):123-32. doi: 10.3109/01674820209042794. PMID 12189897
- [Background] Basson R, Brotto LA. Sexual psychophysiology and effects of sildenafil citrate in oestrogenised women with acquired genital arousal disorder and impaired orgasm: a randomised controlled trial. BJOG. 2003 Nov;110(11):1014-24. PMID 14592587
- See also: primary investigator's website — https://www.directory.ubc.ca/index.cfm?page=personDetail&row=899750943